CLINICAL TRIAL: NCT00848003
Title: Safety of BB-12 Supplemented Strawberry Yogurt For Healthy Adults on Antibiotics
Acronym: PHASE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Merenstein, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R21AT003600-01A1; IND # 13691 (Other: FDA)
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Adults on Antibiotics
Keywords: Probiotics; BB-12; Yogurt; Antibiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Active (Active Comparator): Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12 (BB-12)
  Probiotic, BB-12, supplemented yogurt, 4 ounces taken orally for 10 days
  Interventions: Drug: Bifidobacterium animalis subsp. lactis strain BB-12
- 2. Placebo (Placebo Comparator): Strawberry flavored yogurt
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bifidobacterium animalis subsp. lactis strain BB-12 — Bifidobacterium animalis subsp. lactis (B. lactis) strain BB-12 (BB-12) probiotic supplemented yogurt, 4 ounces taken orally for 10 days
  Other Names: BB-12 probiotic supplemented yogurt
  Arms: 1. Active
Drug: Placebo — Strawberry flavored yogurt
  Other Names: Strawberry flavored yogurt
  Arms: 2. Placebo

SUMMARY:
We believe a readily available drink containing a high dose of probiotics has the potential to improve compliance through many of these mechanisms. This product also has the potential to positively impact the health of children and adults around the world, as yogurt will likely be more appealing to both children and their parents for long term consumption than pharmaceutical-like preparations. In addition to the benefits associated with the consumption of probiotics, there is an increased health benefit from consuming yogurt, a nutrient dense food.

More specifically, the rationale for this Phase I study is to determine safety of our drink and comply with the FDA's recommendations pertaining to an IND application, we will conduct a phase I safety study.

We hypothesize that BB-12 is safe in healthy adults ages 18 and over.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and write English or Spanish
* Refrigerator for proper storage of drink
* Telephone access
* Enrollment must take place within 24 hours of starting antibiotics
* Treatment with a penicillin class antibiotic regimen for 10 days for an upper respiratory infection;

The following is a list of inclusive antibiotics:

1. Amoxicillin
2. Augmentin (amoxicillin/clavulanate)
3. Ancef (cefazolin)
4. Cefadroxil
5. Cephalexin
6. Cephradine
7. Duricef (cefadroxil)
8. Keflex (cephalexin)
9. Kefzol (cefazolin)
10. Velosef (cephradine)
11. Ceclor (cefaclor)
12. Cefotan
13. Cefoxitin
14. Ceftin (cefuroxime)
15. Cefzil (cefprozil)
16. Lorabid (loracarbef)
17. Mefoxin (Cefoxitin)
18. Zinacef (cefuroxime)
19. Omnicef (cefdinir)
20. Suprax (cefixime)
21. Dicloxacillin
22. Pen-Vee K (penicillin)

    * Antibiotic prescribed at least twice a day
    * Outpatients

Exclusion Criteria:

* Chronic conditions, such as diabetes or asthma, that require daily medication
* Allergy to strawberry
* Active diarrhea
* Allergy to penicillin class antibiotic
* Any other medicines used except prescribed antibiotic and anti-pyretic medicines
* Allergy to any of the following medications

  1. Tetracycline
  2. Erythromycin
  3. Trimethoprim
  4. Ciprofloxacin
* Lactose intolerance.
* During baseline physical exam, any of the following will be grounds for exclusion; systolic blood pressure>140, systolic blood pressure <90, diastolic >90, oxygen saturation <98%, pulse rate >100, pulse rate <55 and respiratory rate >17. These include all vital signs that fall outside of the "normal" range, including Grade 1 through Grade 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to assess the safety of BB-12 yogurt when consumed by generally healthy adults who are consuming antibiotics. | 1 year

SECONDARY OUTCOMES:
In addition to safety diary, participants will keep a daily diary to track number of bowel movements, if drink was consumed, if illness resulted in change in activity, over-the-counter medicines used and other illness symptoms. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Heath and Nutritional Properties of Probiotics in Food Including Powder Milk With Live Lactic Acid Bacteria: Food and Agriculture Organization of the United Nations and World Health Organization2005; 2001.
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Lin HC, Su BH, Chen AC, Lin TW, Tsai CH, Yeh TF, Oh W. Oral probiotics reduce the incidence and severity of necrotizing enterocolitis in very low birth weight infants. Pediatrics. 2005 Jan;115(1):1-4. doi: 10.1542/peds.2004-1463. PMID 15629973
- [Background] Mastrandrea F, Coradduzza G, Serio G, Minardi A, Manelli M, Ardito S, Muratore L. Probiotics reduce the CD34+ hemopoietic precursor cell increased traffic in allergic subjects. Eur Ann Allergy Clin Immunol. 2004 Apr;36(4):118-22. PMID 15180351
- [Background] Rosenfeldt V, Michaelsen KF, Jakobsen M, Larsen CN, Moller PL, Pedersen P, Tvede M, Weyrehter H, Valerius NH, Paerregaard A. Effect of probiotic Lactobacillus strains in young children hospitalized with acute diarrhea. Pediatr Infect Dis J. 2002 May;21(5):411-6. doi: 10.1097/00006454-200205000-00012. PMID 12150178
- [Background] Vanderhoof JA, Whitney DB, Antonson DL, Hanner TL, Lupo JV, Young RJ. Lactobacillus GG in the prevention of antibiotic-associated diarrhea in children. J Pediatr. 1999 Nov;135(5):564-8. doi: 10.1016/s0022-3476(99)70053-3. PMID 10547243
- [Background] Pelletier S, Kundrat S, Hasler CM. Effects of a functional foods nutrition education program with cardiac rehabilitation patients. J Cardiopulm Rehabil. 2003 Sep-Oct;23(5):334-40. doi: 10.1097/00008483-200309000-00002. PMID 14512777
- [Background] Pelletier S, Kundrat S, Hasler CM. Effects of an educational program on intent to consume functional foods. J Am Diet Assoc. 2002 Sep;102(9):1297-300. doi: 10.1016/s0002-8223(02)90286-5. PMID 12792631
- [Background] Hasler CM, Bloch AS, Thomson CA, Enrione E, Manning C. Position of the American Dietetic Association: Functional foods. J Am Diet Assoc. 2004 May;104(5):814-26. doi: 10.1016/j.jada.2004.03.015. PMID 15127071
- [Background] Van den Driessche M, Veereman-Wauters G. Functional foods in pediatrics. Acta Gastroenterol Belg. 2002 Jan-Mar;65(1):45-51. PMID 12014316
- [Background] Research MM. The Live Active Culture Yogurt Survey. Monroe Mendelsohn Research. Available at: http://www.dannon.com/dn/dnstore/cgi-bin/ProdDetEv_Cat_240861_SubCat_240857_NavRoot_200_NavID_241709_ProdID_289256.htm. Accessed May 24, 2005.
- [Background] Tuohy KM, Rouzaud GC, Bruck WM, Gibson GR. Modulation of the human gut microflora towards improved health using prebiotics--assessment of efficacy. Curr Pharm Des. 2005;11(1):75-90. doi: 10.2174/1381612053382331. PMID 15638753
- [Background] Veilleux BG, Rowland I. Simulation of the rat intestinal ecosystem using a two-stage continuous culture system. J Gen Microbiol. 1981 Mar;123(1):103-15. doi: 10.1099/00221287-123-1-103. PMID 7033452
- [Background] Clausen MR, Bonnen H, Tvede M, Mortensen PB. Colonic fermentation to short-chain fatty acids is decreased in antibiotic-associated diarrhea. Gastroenterology. 1991 Dec;101(6):1497-504. doi: 10.1016/0016-5085(91)90384-w. PMID 1955116
- [Background] Engelbrektson AL, Korzenik JR, Sanders ME, Clement BG, Leyer G, Klaenhammer TR, Kitts CL. Analysis of treatment effects on the microbial ecology of the human intestine. FEMS Microbiol Ecol. 2006 Aug;57(2):239-50. doi: 10.1111/j.1574-6941.2006.00112.x. PMID 16867142
- [Background] Klijn A, Mercenier A, Arigoni F. Lessons from the genomes of bifidobacteria. FEMS Microbiol Rev. 2005 Aug;29(3):491-509. doi: 10.1016/j.femsre.2005.04.010. PMID 15939502
- [Background] Langhendries JP, Detry J, Van Hees J, Lamboray JM, Darimont J, Mozin MJ, Secretin MC, Senterre J. Effect of a fermented infant formula containing viable bifidobacteria on the fecal flora composition and pH of healthy full-term infants. J Pediatr Gastroenterol Nutr. 1995 Aug;21(2):177-81. doi: 10.1097/00005176-199508000-00009. PMID 7472904
- [Background] Meile L, Ludwig W, Rueger U, et al. Bifidobacterium lactis sp. nov., a moderately oxygen tolerant species isolated from fermented milk. Syst. Appl. Microbiol. 1997(20):57-46.
- [Background] Fuller R. Probiotics in human medicine. Gut. 1991 Apr;32(4):439-42. doi: 10.1136/gut.32.4.439. No abstract available. PMID 1902810
- [Background] Perdigon G, de Macias ME, Alvarez S, Oliver G, de Ruiz Holgado AA. Effect of perorally administered lactobacilli on macrophage activation in mice. Infect Immun. 1986 Aug;53(2):404-10. doi: 10.1128/iai.53.2.404-410.1986. PMID 3733223
- [Background] Wilson KH, Perini F. Role of competition for nutrients in suppression of Clostridium difficile by the colonic microflora. Infect Immun. 1988 Oct;56(10):2610-4. doi: 10.1128/iai.56.10.2610-2614.1988. PMID 3417352
- [Background] Pongpech P, Hentges DJ, Marsh WW, Eberle ME. Effect of streptomycin administration on association of enteric pathogens with cecal tissue of mice. Infect Immun. 1989 Jul;57(7):2092-7. doi: 10.1128/iai.57.7.2092-2097.1989. PMID 2659535
- [Background] Sartor RB. Probiotic therapy of intestinal inflammation and infections. Curr Opin Gastroenterol. 2005 Jan;21(1):44-50. PMID 15687884
- [Background] Sartor RB. Therapeutic manipulation of the enteric microflora in inflammatory bowel diseases: antibiotics, probiotics, and prebiotics. Gastroenterology. 2004 May;126(6):1620-33. doi: 10.1053/j.gastro.2004.03.024. PMID 15168372
- [Background] Davidson JN, Hirsh DC. Bacterial competition as a means of preventing neonatal diarrhea in pigs. Infect Immun. 1976 Jun;13(6):1773-4. doi: 10.1128/iai.13.6.1773-1774.1976. PMID 786883
- [Background] Cong Y, Konrad A, Iqbal N, Elson CO. Probiotics and immune regulation of inflammatory bowel diseases. Curr Drug Targets Inflamm Allergy. 2003 Jun;2(2):145-54. doi: 10.2174/1568010033484278. PMID 14561167
- [Background] Rautava S, Kalliomaki M, Isolauri E. Probiotics during pregnancy and breast-feeding might confer immunomodulatory protection against atopic disease in the infant. J Allergy Clin Immunol. 2002 Jan;109(1):119-21. doi: 10.1067/mai.2002.120273. PMID 11799376
- [Background] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Background] Jijon H, Backer J, Diaz H, Yeung H, Thiel D, McKaigney C, De Simone C, Madsen K. DNA from probiotic bacteria modulates murine and human epithelial and immune function. Gastroenterology. 2004 May;126(5):1358-73. doi: 10.1053/j.gastro.2004.02.003. PMID 15131797
- [Background] Kruis W, Fric P, Pokrotnieks J, Lukas M, Fixa B, Kascak M, Kamm MA, Weismueller J, Beglinger C, Stolte M, Wolff C, Schulze J. Maintaining remission of ulcerative colitis with the probiotic Escherichia coli Nissle 1917 is as effective as with standard mesalazine. Gut. 2004 Nov;53(11):1617-23. doi: 10.1136/gut.2003.037747. PMID 15479682
- [Background] Kruis W, Schutz E, Fric P, Fixa B, Judmaier G, Stolte M. Double-blind comparison of an oral Escherichia coli preparation and mesalazine in maintaining remission of ulcerative colitis. Aliment Pharmacol Ther. 1997 Oct;11(5):853-8. doi: 10.1046/j.1365-2036.1997.00225.x. PMID 9354192
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Gionchetti P, Rizzello F, Venturi A, Brigidi P, Matteuzzi D, Bazzocchi G, Poggioli G, Miglioli M, Campieri M. Oral bacteriotherapy as maintenance treatment in patients with chronic pouchitis: a double-blind, placebo-controlled trial. Gastroenterology. 2000 Aug;119(2):305-9. doi: 10.1053/gast.2000.9370. PMID 10930365
- [Background] Rembacken BJ, Snelling AM, Hawkey PM, Chalmers DM, Axon AT. Non-pathogenic Escherichia coli versus mesalazine for the treatment of ulcerative colitis: a randomised trial. Lancet. 1999 Aug 21;354(9179):635-9. doi: 10.1016/s0140-6736(98)06343-0. PMID 10466665
- [Background] Fukushima Y, Kawata Y, Hara H, Terada A, Mitsuoka T. Effect of a probiotic formula on intestinal immunoglobulin A production in healthy children. Int J Food Microbiol. 1998 Jun 30;42(1-2):39-44. doi: 10.1016/s0168-1605(98)00056-7. PMID 9706796
- [Background] Fukushima Y, Kwata Y, H H. Effect of a probiotic formula containing bifidobacteria (Nan BF) on fecal flora and fecal metaboiltes in healthy children. Bioscience Microflora. 1997(16):65-72.
- [Background] Malinen E, Matto J, Salmitie M, Alander M, Saarela M, Palva A. PCR-ELISA II: Analysis of Bifidobacterium populations in human faecal samples from a consumption trial with Bifidobacterium lactis Bb-12 and a galacto-oligosaccharide preparation. Syst Appl Microbiol. 2002 Aug;25(2):249-58. doi: 10.1078/0723-2020-00117. PMID 12353880
- [Background] Ouwehand AC, Kurvinen T, Rissanen P. Use of a probiotic Bifidobacterium in a dry food matrix, an in vivo study. Int J Food Microbiol. 2004 Aug 15;95(1):103-6. doi: 10.1016/j.ijfoodmicro.2004.03.015. PMID 15240080
- [Background] Bartosch S, Woodmansey EJ, Paterson JC, McMurdo ME, Macfarlane GT. Microbiological effects of consuming a synbiotic containing Bifidobacterium bifidum, Bifidobacterium lactis, and oligofructose in elderly persons, determined by real-time polymerase chain reaction and counting of viable bacteria. Clin Infect Dis. 2005 Jan 1;40(1):28-37. doi: 10.1086/426027. Epub 2004 Dec 6. PMID 15614689
- [Background] Salminen S, von Wright A, Morelli L, Marteau P, Brassart D, de Vos WM, Fonden R, Saxelin M, Collins K, Mogensen G, Birkeland SE, Mattila-Sandholm T. Demonstration of safety of probiotics -- a review. Int J Food Microbiol. 1998 Oct 20;44(1-2):93-106. doi: 10.1016/s0168-1605(98)00128-7. PMID 9849787
- [Background] Turck D, Bernet JP, Marx J, Kempf H, Giard P, Walbaum O, Lacombe A, Rembert F, Toursel F, Bernasconi P, Gottrand F, McFarland LV, Bloch K. Incidence and risk factors of oral antibiotic-associated diarrhea in an outpatient pediatric population. J Pediatr Gastroenterol Nutr. 2003 Jul;37(1):22-6. doi: 10.1097/00005176-200307000-00004. PMID 12827001
- [Background] Mitchell DK, Van R, Mason EH, Norris DM, Pickering LK. Prospective study of toxigenic Clostridium difficile in children given amoxicillin/clavulanate for otitis media. Pediatr Infect Dis J. 1996 Jun;15(6):514-9. doi: 10.1097/00006454-199606000-00008. PMID 8783348
- [Background] McCarty JM, Phillips A, Wiisanen R. Comparative safety and efficacy of clarithromycin and amoxicillin/clavulanate in the treatment of acute otitis media in children. Pediatr Infect Dis J. 1993 Dec;12(12 Suppl 3):S122-7. doi: 10.1097/00006454-199312003-00006. PMID 8295813
- [Background] Elstner CL, Lindsay AN, Book LS, Matsen JM. Lack of relationship of Clostridium difficile to antibiotic-associated diarrhea in children. Pediatr Infect Dis. 1983 Sep-Oct;2(5):364-6. doi: 10.1097/00006454-198309000-00006. PMID 6634465
- [Background] McFarland LV. Epidemiology, risk factors and treatments for antibiotic-associated diarrhea. Dig Dis. 1998 Sep-Oct;16(5):292-307. doi: 10.1159/000016879. PMID 9892789
- [Background] Beaugerie L, Flahault A, Barbut F, Atlan P, Lalande V, Cousin P, Cadilhac M, Petit JC; Study Group. Antibiotic-associated diarrhoea and Clostridium difficile in the community. Aliment Pharmacol Ther. 2003 Apr 1;17(7):905-12. doi: 10.1046/j.1365-2036.2003.01531.x. PMID 12656693
- [Background] Young VB, Schmidt TM. Antibiotic-associated diarrhea accompanied by large-scale alterations in the composition of the fecal microbiota. J Clin Microbiol. 2004 Mar;42(3):1203-6. doi: 10.1128/JCM.42.3.1203-1206.2004. PMID 15004076
- [Background] Finkelstein JA, Davis RL, Dowell SF, Metlay JP, Soumerai SB, Rifas-Shiman SL, Higham M, Miller Z, Miroshnik I, Pedan A, Platt R. Reducing antibiotic use in children: a randomized trial in 12 practices. Pediatrics. 2001 Jul;108(1):1-7. doi: 10.1542/peds.108.1.1. PMID 11433046
- [Background] Finkelstein JA, Metlay JP, Davis RL, Rifas-Shiman SL, Dowell SF, Platt R. Antimicrobial use in defined populations of infants and young children. Arch Pediatr Adolesc Med. 2000 Apr;154(4):395-400. doi: 10.1001/archpedi.154.4.395. PMID 10768680
- [Background] Nyquist AC, Gonzales R, Steiner JF, Sande MA. Antibiotic prescribing for children with colds, upper respiratory tract infections, and bronchitis. JAMA. 1998 Mar 18;279(11):875-7. doi: 10.1001/jama.279.11.875. PMID 9516004
- [Background] McCaig LF, Hughes JM. Trends in antimicrobial drug prescribing among office-based physicians in the United States. JAMA. 1995 Jan 18;273(3):214-9. PMID 7807660
- [Background] McCaig LF, Besser RE, Hughes JM. Antimicrobial drug prescription in ambulatory care settings, United States, 1992-2000. Emerg Infect Dis. 2003 Apr;9(4):432-7. doi: 10.3201/eid0904.020268. PMID 12702222
- [Background] Stille CJ, Andrade SE, Huang SS, Nordin J, Raebel MA, Go AS, Chan KA, Finkelstein JA. Increased use of second-generation macrolide antibiotics for children in nine health plans in the United States. Pediatrics. 2004 Nov;114(5):1206-11. doi: 10.1542/peds.2004-0311. PMID 15520097
- [Background] Cremonini F, Di Caro S, Nista EC, Bartolozzi F, Capelli G, Gasbarrini G, Gasbarrini A. Meta-analysis: the effect of probiotic administration on antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2002 Aug;16(8):1461-7. doi: 10.1046/j.1365-2036.2002.01318.x. PMID 12182746
- [Background] Szajewska H, Mrukowicz JZ. Use of probiotics in children with acute diarrhea. Paediatr Drugs. 2005;7(2):111-22. doi: 10.2165/00148581-200507020-00004. PMID 15871631
- [Background] Szajewska H, Mrukowicz JZ. Probiotics in prevention of antibiotic-associated diarrhea: meta-analysis. J Pediatr. 2003 Jan;142(1):85. No abstract available. PMID 12569905
- [Background] McFarland LV. Meta-analysis of probiotics for the prevention of antibiotic associated diarrhea and the treatment of Clostridium difficile disease. Am J Gastroenterol. 2006 Apr;101(4):812-22. doi: 10.1111/j.1572-0241.2006.00465.x. PMID 16635227
- [Background] Hawrelak JA, Whitten DL, Myers SP. Is Lactobacillus rhamnosus GG effective in preventing the onset of antibiotic-associated diarrhoea: a systematic review. Digestion. 2005;72(1):51-6. doi: 10.1159/000087637. Epub 2005 Aug 18. PMID 16113542
- [Background] D'Souza AL, Rajkumar C, Cooke J, Bulpitt CJ. Probiotics in prevention of antibiotic associated diarrhoea: meta-analysis. BMJ. 2002 Jun 8;324(7350):1361. doi: 10.1136/bmj.324.7350.1361. PMID 12052801
- [Background] Correa NB, Peret Filho LA, Penna FJ, Lima FM, Nicoli JR. A randomized formula controlled trial of Bifidobacterium lactis and Streptococcus thermophilus for prevention of antibiotic-associated diarrhea in infants. J Clin Gastroenterol. 2005 May-Jun;39(5):385-9. doi: 10.1097/01.mcg.0000159217.47419.5b. PMID 15815206
- [Background] Arvola T, Laiho K, Torkkeli S, Mykkanen H, Salminen S, Maunula L, Isolauri E. Prophylactic Lactobacillus GG reduces antibiotic-associated diarrhea in children with respiratory infections: a randomized study. Pediatrics. 1999 Nov;104(5):e64. doi: 10.1542/peds.104.5.e64. PMID 10545590
- [Background] Kim YI. Will mandatory folic acid fortification prevent or promote cancer? Am J Clin Nutr. 2004 Nov;80(5):1123-8. doi: 10.1093/ajcn/80.5.1123. PMID 15531657
- [Background] Williams LJ, Rasmussen SA, Flores A, Kirby RS, Edmonds LD. Decline in the prevalence of spina bifida and anencephaly by race/ethnicity: 1995-2002. Pediatrics. 2005 Sep;116(3):580-6. doi: 10.1542/peds.2005-0592. PMID 16140696
- [Background] Hasler CM. Functional foods: benefits, concerns and challenges-a position paper from the american council on science and health. J Nutr. 2002 Dec;132(12):3772-81. doi: 10.1093/jn/132.12.3772. PMID 12468622
- [Background] Avery JK. Making the most of cholesterol-lowering margarines. Cleve Clin J Med. 2001 Mar;68(3):194-6. doi: 10.3949/ccjm.68.3.194. PMID 11263847
- [Background] Tammi A, Ronnemaa T, Gylling H, Rask-Nissila L, Viikari J, Tuominen J, Pulkki K, Simell O. Plant stanol ester margarine lowers serum total and low-density lipoprotein cholesterol concentrations of healthy children: the STRIP project. Special Turku Coronary Risk Factors Intervention Project. J Pediatr. 2000 Apr;136(4):503-10. doi: 10.1016/s0022-3476(00)90014-3. PMID 10753249
- [Background] Hasler CM. Functional Foods: Their Role in Diease Prevention and Health Promotion. Food Technology. 1998;52(2):57-62.
- [Background] Hasler CM, Kundrat S, Wool D. Functional foods and cardiovascular disease. Curr Atheroscler Rep. 2000 Nov;2(6):467-75. doi: 10.1007/s11883-000-0045-9. PMID 11122780
- [Background] St-Onge MP. Dietary fats, teas, dairy, and nuts: potential functional foods for weight control? Am J Clin Nutr. 2005 Jan;81(1):7-15. doi: 10.1093/ajcn/81.1.7. PMID 15640454
- [Background] Floch MH, Hong-Curtiss J. Probiotics and Functional Foods in Gastrointestinal Disorders. Curr Treat Options Gastroenterol. 2002 Aug;5(4):311-321. doi: 10.1007/s11938-002-0054-6. PMID 12095479
- [Background] Hamilton-Miller JM, Shah S, Winkler JT. Public health issues arising from microbiological and labelling quality of foods and supplements containing probiotic microorganisms. Public Health Nutr. 1999 Jun;2(2):223-9. doi: 10.1017/s1368980099000282. PMID 10447251
- [Background] Beniwal RS, Arena VC, Thomas L, Narla S, Imperiale TF, Chaudhry RA, Ahmad UA. A randomized trial of yogurt for prevention of antibiotic-associated diarrhea. Dig Dis Sci. 2003 Oct;48(10):2077-82. doi: 10.1023/a:1026155328638. PMID 14627358
- [Background] Alm L, Ryd-Kjellen E, Setterberg G, Blomquist L. Effect of a new fermented milk product
- [Background] Black FT, Anderson PL, Orskov J, Orskov F, Gaarslev K, Laulund S. Prophylactic efficacy of lactobacilli on traveler's diarrhea. Travel Medicine. 1989:333-335.
- [Background] Chouraqui JP, Van Egroo LD, Fichot MC. Acidified milk formula supplemented with bifidobacterium lactis: impact on infant diarrhea in residential care settings. J Pediatr Gastroenterol Nutr. 2004 Mar;38(3):288-92. doi: 10.1097/00005176-200403000-00011. PMID 15076628
- [Background] Saavedra JM, Bauman NA, Oung I, Perman JA, Yolken RH. Feeding of Bifidobacterium bifidum and Streptococcus thermophilus to infants in hospital for prevention of diarrhoea and shedding of rotavirus. Lancet. 1994 Oct 15;344(8929):1046-9. doi: 10.1016/s0140-6736(94)91708-6. PMID 7934445
- [Background] Phuapradit P, Varavithya W, Vathanophas K, Sangchai R, Podhipak A, Suthutvoravut U, Nopchinda S, Chantraruksa V, Haschke F. Reduction of rotavirus infection in children receiving bifidobacteria-supplemented formula. J Med Assoc Thai. 1999 Nov;82 Suppl 1:S43-8. PMID 10730517
- [Background] Schiffrin EJ, Rochat F, Link-Amster H, Aeschlimann JM, Donnet-Hughes A. Immunomodulation of human blood cells following the ingestion of lactic acid bacteria. J Dairy Sci. 1995 Mar;78(3):491-7. doi: 10.3168/jds.S0022-0302(95)76659-0. PMID 7782506
- [Background] Link-Amster H, Rochat F, Saudan KY, Mignot O, Aeschlimann JM. Modulation of a specific humoral immune response and changes in intestinal flora mediated through fermented milk intake. FEMS Immunol Med Microbiol. 1994 Nov;10(1):55-63. doi: 10.1111/j.1574-695X.1994.tb00011.x. PMID 7874079
- [Background] Kankaanpaa P, Sutas Y, Salminen S, Isolauri E. Results on clinical demonstration of probiotics on children. Paper presented at: Presented at Functional Food Research in Europe, Third Workshop, 1998; Probdemo, Finland, October 1-2.
- [Background] Amrouche T, Boutin Y, Fliss I. Effects of bifidobacterial cytoplasm peptide and protein fractions on mouse lymphocyte proliferation and cytokine production. Food and Agricultural Immunology. MAR 2006;17(1):29-42.
- [Background] Amrouche T, Boutin Y, Prioult G, Fliss I. Effects of bifidobacterial cytoplasm, cell wall and exopolysaccharide on mouse lymphocyte proliferation and cytokine production. International Dairy Journal. JAN 2006;16(1):70-80.
- [Background] Matsumoto M, Ohishi H, Benno Y. Impact of LKM512 yogurt on improvement of intestinal environment of the elderly. FEMS Immunol Med Microbiol. 2001 Oct;31(3):181-6. doi: 10.1111/j.1574-695X.2001.tb00518.x. PMID 11720813
- [Background] Obradovic D, Curic M, Ivanovic M, Trbojevic B, Djordjevic M. Probiotic function of the fermented milk Jogurt Plus. Paper presented at: FEMS Conference (Fifthe Symposium on Lactic Acid Bacteria), 1996; Holland. September 8-12.
- [Background] Nord CE, Lidbeck A, Orrhage K, Sjostedt S. Oral supplementation with lactic acid-producing bacteria during intake of clindamycin. Clin Microbiol Infect. 1997 Feb;3(1):124-132. doi: 10.1111/j.1469-0691.1997.tb00262.x. PMID 11864087
- [Background] Salminen S, Laine M, von Wright A, Vuopio-Varkila J, Kohonen T, Mattila-Sandholm T. Development of selection criteria for probiotic strains to assess their potential in functional foods: A Nordic and European approach. Bioscience Microflora. 1996;15(2):61-67.
- [Background] Black FT, Laulund S. A study on the recovery of ingested, encapsulated Lactobacillus acidophilus and Bifidobacteria bifidum from doudenal fluid and faeces. Chr. Hansen Internal Report. 1988.
- [Background] Abi-Hanna A, Moore N, Yolken RH, Saavedra JM. Long term consumption of infant formulas with live probiotic bacteria: safety and tolerance. Journal of Pediatric Gastroenterology and Nutrition. 1998;27(4):484.
- [Background] Saavedra JM, Abi-Hanna A, Moore N, Yolken RH. Long-term consumption of infant formulas containing live probiotic bacteria: tolerance and safety. Am J Clin Nutr. 2004 Feb;79(2):261-7. doi: 10.1093/ajcn/79.2.261. PMID 14749232
- [Background] Lourens-Hattingh A, Viljoen BC. Yogurt as probiotic carrier food. International Dairy Journal. 2001;11(1-2):1-17.
- [Background] Tammam JD, Williams AG, Banks J, Cowie G, Lloyd D. Membrane inlet mass spectrometric measurement of O2 and CO2 gradients in cultures of Lactobacillus paracasei and a developing Cheddar cheese ecosystem. Int J Food Microbiol. 2001 Apr 11;65(1-2):11-22. doi: 10.1016/s0168-1605(00)00438-4. PMID 11322693
- [Background] Gonzales R, Steiner JF, Sande MA. Antibiotic prescribing for adults with colds, upper respiratory tract infections, and bronchitis by ambulatory care physicians. JAMA. 1997 Sep 17;278(11):901-4. PMID 9302241
- [Background] Gill JM, Fleischut P, Haas S, Pellini B, Crawford A, Nash DB. Use of antibiotics for adult upper respiratory infections in outpatient settings: a national ambulatory network study. Fam Med. 2006 May;38(5):349-54. PMID 16673197
- [Background] Steinman MA, Gonzales R, Linder JA, Landefeld CS. Changing use of antibiotics in community-based outpatient practice, 1991-1999. Ann Intern Med. 2003 Apr 1;138(7):525-33. doi: 10.7326/0003-4819-138-7-200304010-00008. PMID 12667022
- [Background] Glass RI, Lew JF, Gangarosa RE, LeBaron CW, Ho MS. Estimates of morbidity and mortality rates for diarrheal diseases in American children. J Pediatr. 1991 Apr;118(4 Pt 2):S27-33. doi: 10.1016/s0022-3476(05)81422-2. PMID 2007954
- [Background] Gangarosa RE, Glass RI, Lew JF, Boring JR. Hospitalizations involving gastroenteritis in the United States, 1985: the special burden of the disease among the elderly. Am J Epidemiol. 1992 Feb 1;135(3):281-90. doi: 10.1093/oxfordjournals.aje.a116282. PMID 1546704
- [Background] Ho MS, Glass RI, Pinsky PF, Young-Okoh NC, Sappenfield WM, Buehler JW, Gunter N, Anderson LJ. Diarrheal deaths in American children. Are they preventable? JAMA. 1988 Dec 9;260(22):3281-5. PMID 3184416
- [Background] Ho MS, Glass RI, Pinsky PF, Anderson LJ. Rotavirus as a cause of diarrheal morbidity and mortality in the United States. J Infect Dis. 1988 Nov;158(5):1112-6. doi: 10.1093/infdis/158.5.1112. No abstract available. PMID 3183422
- [Background] Haynes RB, Yao X, Degani A, Kripalani S, Garg A, McDonald HP. Interventions to enhance medication adherence. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD000011. doi: 10.1002/14651858.CD000011.pub2. PMID 16235271
- [Background] Winnick S, Lucas DO, Hartman AL, Toll D. How do you improve compliance? Pediatrics. 2005 Jun;115(6):e718-24. doi: 10.1542/peds.2004-1133. PMID 15930200
- [Background] Ansah EK, Gyapong JO, Agyepong IA, Evans DB. Improving adherence to malaria treatment for children: the use of pre-packed chloroquine tablets vs. chloroquine syrup. Trop Med Int Health. 2001 Jul;6(7):496-504. doi: 10.1046/j.1365-3156.2001.00740.x. PMID 11469941
- [Background] Nevins TE.